CLINICAL TRIAL: NCT04803682
Title: ASPIRE+ Mentoring Moon Shot Youth Lung Prevention
Brief Title: A Smoking Prevention Program (ASPIRE) and Mentoring for Preventing Smoking Among High School Youths
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0258; NCI-2019-02481 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0258 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-09; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (ASPIRE, mentorship) (Experimental): Participants complete online ASPIRE course over 3.5-4 hours.
  HIGH SCHOOL MENTORS: Eleventh grade high school students receive mentor training over 4-5 hours on how to mentor ninth grade students.
  ALL STUDENTS: Mentors and mentees are paired up so that eleventh grade high school students mentor the ninth grade high school students over 30 minutes for 7 sessions about the different types of tobacco products (such as cigarettes, cigars, hookah, and so on) and the dangers of these products.
  Interventions: Behavioral: Preventive Intervention; Behavioral: Questionnaire Administration

INTERVENTIONS:
Behavioral: Preventive Intervention — Participate in ASPIRE and mentorship program
  Other Names: PREVENTATIVE; Prevention; Prevention Measures; prophylaxis; PRYLX
Behavioral: Questionnaire Administration — Ancillary studies (pre and post questionnaire)

SUMMARY:
This early phase I trial studies how well A Smoking Prevention Interactive Experience (ASPIRE) program and mentorship works in preventing smoking in high school students. ASPIRE is an online-based, youth-centered tobacco prevention and cessation program. The goal of this research study is to learn if training eleventh grade high school students to be tobacco-free role models and mentors for ninth grade high school students is possible and will positively influence the younger peers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of training selected eleventh grade high school student volunteers to provide an intervention involving mentoring combined with social support activities.

II. To increase ninth grade high school student well-being, which would ultimately influence tobacco related knowledge and resistance skills regarding tobacco uptake among ninth grade high school program participants.

EXPLORATORY OBJECTIVES:

I. Mentor ability, confidence, and intention (ACI) to address tobacco use and dependence and providing anti-tobacco advice to mentees.

II. To determine the scores on mentoring competencies. III. To determine the influences of social support and self-esteem by mentors. IV. To determine the quality and satisfaction with the relationships among mentors and mentees.

V. To determine level of knowledge about nicotine and tobacco products among mentees.

VI. To determine susceptibility to tobacco use among non-smokers. VII. To determine progression through stages of change among smokers.

OUTLINE:

Participants complete online ASPIRE course over 3.5-4 hours.

HIGH SCHOOL MENTORS: Eleventh grade high school students receive mentor training over 4-5 hours on how to mentor ninth grade students.

ALL STUDENTS: Mentors and mentees are paired up so that eleventh grade high school students mentor the ninth grade high school students over 30 minutes for 7 sessions about the different types of tobacco products (such as cigarettes, cigars, hookah, and so on) and the dangers of these products.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-18
* Enrolled in grades nine or eleven
* Speaks and understands English
* Parent or legally authorized guardian (LAR) provide written consent for study participation
* Student provides written assent for study participation

Exclusion Criteria

* Unable to speak and understand English
* Lives in the same household with another participant in the study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Required number of participants should be 40 mentors and 100 mentees | 3 years
  At least 40 mentors and 100 mentees.
Number of participants required to complete baseline and post-intervention assessments should be 35 mentors and 80 mentees | 3 years
  At least 80% completion rates.
All participants are required to attend at least 5 of 7 sessions of mentor to mentees interactions | 3 years
  At least 5 of 7 sessions of mentor/mentee interactions
Participants with the ability to provide the level of satisfaction with the program | 3 years
  Training program for mentors and overall program satisfaction. Seventeen-item rating scale (1 = not skilled at all to 7 = extremely skilled) about facets of mentoring.

SECONDARY OUTCOMES:
Tobacco related knowledge among mentees | 3 years
  Assessed by comparing pre and post intervention scores. Three-item rating scale (0 = no ability/confidence/intention to 4 = high ability, confidence, and intention) Nineteen-item scale measuring quality of mentor to mentee relationship. Four point Likert scale (1 = not true at all to 4 = very true) Twenty-five item scale. Multiple choice questions to measure tobacco and nicotine product knowledge developed by ASPIRE study team

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States